CLINICAL TRIAL: NCT05603611
Title: Implementation of the HELIOSTARTM in Real-world Clinical Practice at a High-volume Center - Operator Learning Curve and Procedural Outcome Parameters
Brief Title: Implementation of the HELIOSTARTM in Real-world Clinical Practice at a High-volume Center
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Maura Zylla, Co-Principal Investigator, University Hospital Heidelberg
Other Study IDs: UHHeidelberg_2
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Pulmonary vein isolation — Local electrical isolation of PV ostia to prevent recurrence of AF due to ectopic PV-triggers

SUMMARY:
The HELIOSTARTM catheter (Biosense Webster) is a new technology for pulmonary vein isolation (PVI) in atrial fibrillation (AF), combining radiofrequency (RF)-ablation and 3D-mapping visualization with the concept of "single-shot"-ablation device. This study evaluates the operator learning curve und procedural outcome during implementation of the HELIOSTARTM.

DETAILED DESCRIPTION:
The first patients undergoing PVI by HELIOSTARTM at Heidelberg University Hospital are included in this prospective study. Procedures are performed by an operator proficient in CB-ablation. Procedural outcome was analyzed over the course of increasing experience with the device and in comparison to a previous cohort investigated during implementation of the Arctic FrontTM-cryoballoon (Medtronic).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years, ability to provide informed consent and at least one episode of documented paroxysmal or persistent AF

Exclusion Criteria:

* history of prior AF ablation, left atrial thrombus, suspected irregular PV-anatomy in pre-procedural transesophageal echocardiography (TOE) or contraindication for peri-procedural anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting at Heidelberg University Hospital with an indication for AF ablation via the clinical routine.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedure duration | Day of index procedure, number of minutes
LA dwell time | Day of index procedure, number of minutes
  Minutes
Fluoroscopy duration | Day of index procedure, number of minutes
  Minutes

SECONDARY OUTCOMES:
Short-term AF arrhythmia recurrence | 3 months
  ECG-documented AF
Procedural complications | 3 months
  As diagnosed by physician and documented in written report
Long-term arrhythmia recurrence | 12 months
  ECG-documented AF

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Department of Cardiology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zylla MM, Leiner J, Rahm AK, Hoffmann T, Lugenbiel P, Schweizer P, Mages C, Mereles D, Kieser M, Scholz E, Katus HA, Frey N, Thomas D. Catheter ablation of atrial fibrillation in women with heart failure with preserved ejection fraction. Front Cardiovasc Med. 2024 Nov 11;11:1463815. doi: 10.3389/fcvm.2024.1463815. eCollection 2024. PMID 39588067